CLINICAL TRIAL: NCT05894889
Title: Single Cell Analysis of CXCL13+PD1+ CD8 T Cell in Association With Resistance to Pembrolizumab and Chemotherapy Neoadjuvant/Adjuvant of NSCLC
Brief Title: Pembrolizumab and Chemotherapy Neoadjuvant/Adjuvant of NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Shanghai Pulmonary Hospital, Shanghai, China (Other); Guangdong Provincial People's Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECT2304029302
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Stage IIIB(N2) Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer
Keywords: Early stage NSCLC, neoadjuvant, adjuvant, pembrolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: None(Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + Chemotherapy (Experimental): Non-squamous NSCLC: pembrolizumab 200mg as at least 30-minute IV infusion on Day 1, followed by pemetrexed at a dose of 500mg/m2 IV over 30 minutes or per institutional standard with Carboplatin at a dose of AUC 5 over 120 minutes or per institutional standard, of a 3-week treatment cycle, for up to 4 cycles.
  Squamous NSCLC: pembrolizumab 200mg as at least 30-minute IV infusion on Day 1, followed by nab-paclitaxel at a dose of 135mg/m2 IV over 30 minutes or per institutional standard with Carboplatin at a dose of AUC 5 over 120 minutes or per institutional standard, of a 3-week treatment cycle, for up to 4 cycles. Nab-paclitaxel will also be administered at the dose of 135mg/m2 for over 30 minutes IV infusion or per institutional standard on day 8 of each 3-week treatment cycle.
  Interventions: Biological: Pembrolizumab 200 mg IV infusion

INTERVENTIONS:
Biological: Pembrolizumab 200 mg IV infusion — Biological: Pembrolizumab 200 mg IV infusion
  Drug: nab-paclitaxel IV infusion
  Drug: Carboplatin IV infusion
  Drug: Pemetrexed IV infusion
  Other Names: Drug: nab-paclitaxel IV infusion; Drug: Carboplatin IV infusion; Drug: Pemetrexed IV infusion

SUMMARY:
This study is to evaluate the efficacy and safety of neoadjuvant pembrolizumab plus chemotherapy following by pembrolizumab adjuvant in stage IIA-IIIB (N2) NSCLC participants without sensitizing EGFR/ALK mutation. The study will also investigate the role of CXCL13+PD1+ CD8 T cells in association with pathological response / resistance to neoadjuvant immunotherapy by comparing the proportion of CXCL13+PD1+ CD8 T cells in all CD8 T cells in post-treatment (surgical sample) between MPR group and non-MPR group.

DETAILED DESCRIPTION:
Lung cancer is still the world's leading cancer in terms of mortality. Although the early screening of lung cancer has made great achievements, for example, many lung cancer patients were already in the middle and late stage of lung cancer when they were diagnosed. The majority of patients with resected Stage II and IIIA NSCLC are destined to suffer tumor recurrence despite the administration of standard adjuvant or neoadjuvant therapy. In recent years, neoadjuvant immunotherapy based on PD-1 receptor has provided new opportunities for surgery of locally advanced NSCLC, including the positive results from KEYNOTE-671 and KEYNOTE-091 study. However the mechanism of immunotherapy response and resistance are still less understood.

CXCL13+ PD1+ CD8 T cells demonstrate an exhausted phenotype and have been proposed as a surrogate of tumor antigen-specific T cell, a key subset of tumor-infiltrating immune cells that have successfully recognized and killed tumor cells but kept from continued functioning by immune checkpoints including PD-L1. Research on T cell exhaustion in chronic viral infection has also suggested that T cell exhaustion is a result of chronic antigen stimulation, corroborating with the notion that exhausted T cells inside the tumor microenvironment represents successful tumor immune recognition

Therefore, in this study, we hypothesize that patients with resectable stage IIA-ⅢB(N2) non-small cell lung cancer (NSCLC) without sensitizing EGFR/ALK mutation could benefit from pembrolizumab combined with chemotherapy. Based on the single cell analysis of the pre-treatment and post-treatment samples, we hypothesize that lack of CXCL13+PD1+ T cells is one of the major resistance mechanisms of PD1/PD-L1 blockade.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of [Stage II, IIIA or IIIB(N2) NSCLC (AJCC Version 8)] will be enrolled in this study.

   Note: mixed cellularity tumors are allowed. tumor should be considered resectable in terms of surgeon's determinations before study entry by investigators. Lymph nodes disease are recommended to have pathological confirmation. A PET-CT may be utilized as a surrogate for pathologic staging by site's feasibility.
2. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 1 year after the last dose of study treatment and refrain from donating sperm during this period.
3. Female participants:

   A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:
   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least [180 days after the last dose of carboplatin and for at least 120 days after the last dose of pembrolizumab, whichever occurs latest].
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial and may also provide consent for future biomedical research.
5. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Participants suspected with secondary lung cancer (eg. ground glass nodules) were also eligible for this study (For solid nodules, biopsy, if available, should be performed in case of any intrapulmonary metastasis).
6. Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
8. Have adequate organ function as defined in the following table. Specimens must be collected within 10 days prior to the start of study intervention.

Exclusion Criteria:

1. Have confirmed sensitizing EGFR mutation or ALK alterations. Note: EGFR and ALK testing will be performed in local hospital, and do not need to be sent to the central laboratory.
2. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
3. Has one of the following tumor locations/types:

   * NSCLC involving the superior sulcus
   * Large cell neuro-endocrine cancer
   * Sarcomatoid tumor
4. Has had an allogenic tissue/solid organ transplant.
5. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
6. Has received prior systemic anti-cancer therapy including investigational agents for the current malignancy prior to [allocation].
7. Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids.
8. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.

   Note: please refer to Section 5.5.2 for information on COVID-19 vaccines
9. Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
12. Has a known severe hypersensitivity (≥Grade 3) to any of the study chemotherapy agents and/or to any of their excipients.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
14. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
15. Has an active infection requiring systemic therapy.
16. Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority.
17. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: Hepatitis B and C screening tests are not required unless:
    * Known history of HBV and HCV infection
    * As mandated by local health authority
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
21. Participants who have had major surgery within 14 days of first treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | Up to approximately 16 months
  pCR in eligible stage IIA-IIIB (N2) NSCLC participants (AJCC Version 8, no known sensitizing EGFR or ALK alterations) following neoadjuvant pembrolizumab plus chemotherapy
Post-treatment proportion of CXCL13+PD1+ CD8 T cells in all CD8 T cells | Up to approximately 16 months
  Post-treatment proportion of CXCL13+PD1+ CD8 T cells in all CD8 T cells in single cell RNA-seq data

SECONDARY OUTCOMES:
MPR in eligible stage IIA-IIIB (N2) NSCLC participants (AJCC Version 8, no known sensitizing EGFR or ALK alterations) following neoadjuvant pembrolizumab plus chemotherapy | Up to approximately 16 months
  MPR rate evaluated by investigator based on protocol defined criteria (the proportion of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes).
Event-free survival (EFS) | Up to approximately 46 months
  EFS is defined as the time from study intervention to the first of the following events:
  * Radiographic disease progression per RECIST 1.1 (for participants who have not had or will not have surgery, participants who have gross residual disease after an incomplete resection [R2 resection]);
  * Local progression (primary tumor or regional lymph nodes) precluding planned surgery;
  * Inability to resect the tumor;
  * Local or distant recurrence (for participants who are disease free after surgery or participants with microscopic positive margins [R1 resection]);
  * Death due to any cause.
Number of Participants with One or More Adverse Events | Up to approximately 46 months
  Participant experiencing AEs, participant discontinuing study intervention due to AEs, and participant experiencing perioperative complications.
PD-L1 TPS(Tumor Proportion Score) evaluation in pre-treatment patients | Up to approximately 16 months
  PD-L1 TPS(Tumor Proportion Score) evaluation in pre-treatment patients of pre-treatment tumor biopsy

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University, Beijing, Beijing Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No